CLINICAL TRIAL: NCT00407797
Title: Pregabalin In Partial Seizures (PREPS): An Open-Label, Multicenter Add On Therapy Trial. A Phase IV Open-Label Trial Using 150,300, 600 mg/Day Of Pregabalin
Brief Title: Pregabalin In Partial Seizures (PREPS): An Open-Label, Multicenter Add On Therapy Trial
Acronym: PREPS MEXICO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081090
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2011-02

CONDITIONS: Partial Seizures
Keywords: Lyrica; Epilepsies - Partial
MeSH Terms: conditions — Seizures; Epilepsies, Partial | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — 150 to 600 mg/day during 21 weeks

SUMMARY:
The purpose of this study is to assess the clinical improvement by partial seizures reduction, safety and tolerability of subjects having partial epilepsy related to the adjunction of pregabalin BID (75 to 300mg day titration, BID) to existing standard AED (Antiepileptic drugs).

DETAILED DESCRIPTION:
This study was terminated on 17 March 2009 due to delayed enrollment. The decision to terminate the trial was not based on any safety concerns, but rather on timelines and the difficulty in enrolling patients in this open label, single group study.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female who are diagnosed of partial seizure (simple partial, complex partial, partial seizure secondarily generalized) as defined in the international league of epilepsy classification of seizure.

Exclusion Criteria:

* Patients having a treatable cause of seizure, currently receiving vigabatrin, having a progressive neurological or systemic disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Mexico (7):
  - Pfizer Investigational Site, México, D. F.
  - Pfizer Investigational Site, Acapulco de Juárez, Guerrero
  - Pfizer Investigational Site, Morelia, Michoacán
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, Aguascalientes
  - Pfizer Investigational Site, Chihuahua City
  - Pfizer Investigational Site, Estado de México

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 152 subjects were screened and 136 subjects were assigned to study treatment.
Groups:
- Pregabalin: 150 mg per day as two doses (75 mg twice daily; BID), increased to 600 mg per day (300 mg BID) as needed based on response and tolerability
Period: Overall Study
Arm/Group | Pregabalin
Started | 136
Full Analysis Set | 135 (At least 1 dose of study medication and had a baseline and at least 1 post-baseline measurement.)
Completed | 118
Not Completed | 18
Not completed — Lost to Follow-up | 2
Not completed — Adverse Event | 6
Not completed — Other | 7
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 136
Age, Customized [Number; unit: participants]
  18 - 44 years | 107
  45 - 64 years | 25
  >= 65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 60
28-Day Seizure Rate [Mean (Standard Deviation); unit: seizure rate] — Number of partial seizures in baseline period divided by duration of period based on observed visit dates multiplied by 28.
  seizure rate | 7.8 (14.0)
28 day seizure frequency in Subjects with <= 6 and > 6 seizures during Baseline Period [Mean (Standard Deviation); unit: seizures] — Baseline period = 8 week period before Visit 1 date, including any unplanned readings falling under this period.
  seizures
    <=6 seizures | 2 (0.8)
    > 6 seizures | 12 (17.2)
Medical Outcomes Study Sleep Scale [Mean (Standard Deviation); unit: scores on scale] — Subject rated questionnaire to assess sleep quality and quantity. For 5 of 7 subscales transformed total score range = 0 to 100; other subscales: Sleep Quantity range: 0-24 hours; and Optimal Sleep range: 1 (optimal sleep: quantity 7 or 8 hours per night), or 0 (no optimal sleep). Higher score indicates greater intensity or quantity of attribute.
  scores on scale
    Sleep Disturbance | 32.9 (20.9)
    Snoring | 40.1 (33.4)
    Awaken Short of Breath | 26.0 (24.8)
    Quantity of Sleep | 7.9 (1.9)
    Optimal Sleep | 0.5 (0.5)
    Sleep Adequacy | 64.6 (26.1)
    Somnolence | 39.2 (24.5)
    9-Item Sleep Problems Index | 33.4 (15.8)
Hospital Anxiety and Depression Scale (HADS) [Mean (Standard Deviation); unit: score on scale] — HADS-A: generalized anxiety; HADS-D: lost interest and diminished pleasure response (lowering of hedonic tone). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
  score on scale
    Anxiety Total Score | 8.8 (4.2)
    Depression Total Score | 7.3 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in 28 Day Partial Seizure Rate During Treatment Observation Phase
Description: 28-day seizure rate (at observation period [obs]) = [(number of seizures obs ) divided by (duration of period based on observed last dosing date and Visit 3 [Week 9] date)] * 28. Percent change = [(28-day seizure rate obs minus 28-day seizure rate at baseline [b]) divided by 28-day seizure rate b] * 100. Negative values indicate a decrease in seizure frequency and positive values reflect an increase in seizure frequency.
Time Frame: Week 9 to Week 21 or End of Treatment (early termination)
Population: Full Analysis Set (FAS): all subjects who received at least 1 dose of assigned treatment, had valid baseline seizure data, and had at least 1 subsequent rating of seizure frequency (modified intent to treat population). N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Pregabalin: 75 mg BID (twice daily); may have been increased to 150 mg BID after Week 1, and to 300 mg BID after Week 2 based on response and tolerability
Arm/Group | Pregabalin
Number analyzed (Participants) | 121
percent change | -51.2 (45.2)
Statistical Analysis 1: Comparison: Pregabalin; Percent change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p < .0001, t-test, 2 sided

2. Secondary Outcome: Response Ratio (RR)
Description: Response ratio (RR) = comparison between baseline 28-seizure frequency with the 12 week observation phase. RR = [(28-day seizure rate in observation period [obs] minus 28-day seizure rate at baseline [b] ) divided by (28-day seizure rate obs plus 28-day seizure rate b)] * 100. Range: -100 to 100; negative values for the RR indicate reductions in seizures.
Time Frame: Week 9 to Week 21 or End of Treatment (early termination)
Population: FAS. N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pregabalin
Number analyzed (Participants) | 121
ratio | -45.1 (37.9)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < .0001, t-test, 2 sided

3. Secondary Outcome: Percent Change From Baseline in 28-Day Partial Seizure Frequency at Week 21
Description: Percent change from Baseline = [(28-day seizure rate at 21 weeks minus 28-day seizure rate at baseline [b]) divided by (28-day seizure rate b) * 100. Negative values indicate a decrease in seizure frequency, positive values reflect an increase in seizure frequency.
Time Frame: Week 21 or End of Treatment (early termination)
Population: FAS.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pregabalin
Number analyzed (Participants) | 135
percent change | -36.0 (55.8)
Statistical Analysis 1: Comparison: Pregabalin; Percent change evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p < .0001, t-test, 2 sided

4. Secondary Outcome: Percent Change From Baseline in Seizure Frequency in Participants Who Had <=6 Seizures and >6 Seizures During the Baseline Period
Description: Negative values indicate a decrease in seizure frequency; positive values reflect an increase in seizure frequency.
Time Frame: Week 9 to Week 21 or End of Treatment (early termination)
Population: FAS. N=number of subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pregabalin
Number analyzed (Participants) | 121
percent change
  <= 6 seizures at Baseline (n=50) | -57.9 (44.9)
  > 6 seizures at Baseline (n=71) | -46.5 (45.1)
Statistical Analysis 1: Comparison: Pregabalin; Participants with <= 6 seizures during Baseline period; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Pregabalin; Participants with > 6 seizures during Baseline Period; Test type: Superiority or Other; p < .0001, t-test, 2 sided

5. Secondary Outcome: Percent of Seizure- Free Participants During the Treatment Observation Period
Description: Seizure-free = no seizures during observation period (100 percent reduction in seizures from baseline).
Time Frame: Week 9 to Week 21 or Early Termination (end of treatment)
Population: FAS. N=number of subjects with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 121
percent of participants | 20.7

6. Secondary Outcome: Percent of Seizure Free Participants During the Last 4 Weeks of the Treatment Observation Period
Description: Seizure-free = no seizures during last 4 weeks of observation period (100 percent reduction in seizures from baseline).
Time Frame: Week 17 to Week 21 (or Last 4 Weeks of Treatment after Week 9)
Population: FAS. N=number of subjects with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 121
percent of participants | 40.5

7. Secondary Outcome: Percent of Participants With >=50% Reduction in Seizure Frequency (28-day Seizure Rate) Between Baseline and Final 4 Weeks of the Treatment Observation Period
Time Frame: Week 17 to Week 21 (or Last 4 Weeks of Treatment after Week 9)
Population: FAS. N=number of subjects with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 121
percent of participants | 63.6

8. Secondary Outcome: Percent of Participants With >=75% Reduction in Seizure Frequency (28-day Seizure Rate) Between Baseline and Final 4 Weeks of the Treatment Observation Period
Time Frame: Week 17 through Week 21 (or Last 4 Weeks of Treatment after Week 9)
Population: FAS. N=number of subjects with evaluable data.
Measure: Number; unit: percent of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 121
percent of participants | 48.8

9. Secondary Outcome: Treatment Satisfaction: Patient General Impression to Change (PGIC)
Description: Patient General Impression to Change (PGIC): participant rated instrument to measure participant's change in overall status since beginning study medication on a 7-point scale; range: 1 (very much improved) to 7 (very much worse). Not done = participant did not complete the PGIC.
Time Frame: Week 21, LOCF
Population: FAS. LOCF = Last Observation Carried Forward.
Measure: Number; unit: percent of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 135
percent of participants
  Week 21: Very Much Improved | 22.4
  Week 21: Much Improved | 52.6
  Week 21: Minimally Improved | 13.8
  Week 21: No Change | 4.3
  Week 21: Minimally Worse | 1.7
  Week 21: Much Worse | 1.7
  Week 21: Very Much Worse | 0.9
  Week 21: Not Done | 2.6
  LOCF: Very Much Improved | 20.7
  LOCF: Much Improved | 51.1
  LOCF: Minimally Improved | 12.6
  LOCF: No Change | 4.4
  LOCF: Minimally Worse | 1.5
  LOCF: Much Worse | 1.5
  LOCF: Very Much Worse | 0.7
  LOCF: Not Done | 7.4

10. Secondary Outcome: Change From Baseline in Sleep Interference: Medical Outcome Sleep Scale (MOS)
Description: Participant rated questionnaire to assess sleep quality and quantity; 9-item overall sleep problems index and 7 subscales. Sleep disturbance, snoring, awaken short of breath, somnolence, and adequacy subscale scores (s) rated 1 (all the time) to 6 (none of the time); transformed s; total range (r): 0 to 100; higher s = greater intensity of attribute; negative values (v) = reduction from baseline (b), positive v = increase from b. Sleep Quantity score r: 0-24 hours. Higher s = greater quantity of sleep. Change = (MOS score at observation period minus MOS score at b) divided by MOS score b.
Time Frame: Week 21, LOCF
Population: FAS. LOCF = Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 135
scores on scale
  Week 21: Sleep Disturbance | -3.8 (20.9)
  LOCF: Sleep Disturbance | -4.0 (21.1)
  Week 21: Snoring | 1.4 (35.4)
  LOCF: Snoring | 2.2 (34.3)
  Week 21: Awaken Short of Breath | 0.7 (32.4)
  LOCF: Awaken Short of Breath | 0.3 (30.9)
  Week 21: Adequacy | 4.2 (28.0)
  LOCF: Adequacy | 4.0 (26.9)
  Week 21: Somnolence | 0.4 (28.3)
  LOCF: Somnolence | -0.8 (28.2)
  Week 21: 9-Item Overall Sleep Problem Index | -2.2 (16.6)
  LOCF: 9-Item Overall Sleep Problem Index | -2.5 (16.1)
  Week 21: Sleep Quantity | 0.4 (2.1)
  LOCF: Sleep Quantity | 0.4 (2.1)
Statistical Analysis 1: Comparison: Pregabalin; Week 21: Sleep Disturbance. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.0552, t-test, 2 sided
Statistical Analysis 2: Comparison: Pregabalin; LOCF: Sleep Disturbance. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.0350, t-test, 2 sided
Statistical Analysis 3: Comparison: Pregabalin; Week 21: Snoring. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.6743, t-test, 2 sided
Statistical Analysis 4: Comparison: Pregabalin; LOCF: Snoring. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.4736, t-test, 2 sided
Statistical Analysis 5: Comparison: Pregabalin; Week 21: Awaken Short of Breath. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.8173, t-test, 2 sided
Statistical Analysis 6: Comparison: Pregabalin; LOCF: Awaken Short of Breath. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.9092, t-test, 2 sided
Statistical Analysis 7: Comparison: Pregabalin; Week 21: Sleep Adequacy. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.1091, t-test, 2 sided
Statistical Analysis 8: Comparison: Pregabalin; LOCF: Sleep Adequacy. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.0944, t-test, 2 sided
Statistical Analysis 9: Comparison: Pregabalin; Week 21: Somnolence. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.8928, t-test, 2 sided
Statistical Analysis 10: Comparison: Pregabalin; LOCF: Somnolence. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.7669, t-test, 2 sided
Statistical Analysis 11: Comparison: Pregabalin; Week 21: 9-Item Overall Sleep Problems Index. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.1698, t-test, 2 sided
Statistical Analysis 12: Comparison: Pregabalin; LOCF: 9-Item Overall Sleep Problem Index. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.0898, t-test, 2 sided
Statistical Analysis 13: Comparison: Pregabalin; Week 21: Quantity of Sleep. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.0465, t-test, 2 sided
Statistical Analysis 14: Comparison: Pregabalin; LOCF: Quantity of Sleep. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.0316, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Sleep Interference: Medical Outcome Sleep Scale (MOS): Optimal Sleep Subscale
Description: Optimal Sleep subscale of the MOS subject rated questionnaire to assess sleep quality and quantity. Optimal Sleep (1 of 7 subscales) was derived from sleep quantity: average hours of sleep each night during the past week. Number of subjects with response: YES=1 (optimal sleep: quantity of sleep was 7 or 8 hours per night) or No= 0 (no optimal sleep). Negative value indicates a decrease in attribute; positive value indicates an increase in attribute. Change = (MOS score at observation period minus MOS score at baseline [b]) divided by MOS score b.
Time Frame: Week 21, LOCF
Population: FAS. LOCF=Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 135
scores on scale
  Week 21 | 0.1 (0.6)
  LOCF | 0.1 (0.6)
Statistical Analysis 1: Comparison: Pregabalin; Week 21; change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.2187, t-test, 2 sided
Statistical Analysis 2: Comparison: Pregabalin; LOCF; change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.1905, t-test, 2 sided

12. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS)
Description: Participant rated questionnaire with 2 subscales: HADS-A assesses generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D: state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale has 7 items; range: 0 (no anxiety or depression) to 3 (severe anxiety or depression). Total score 0 to 21 for each subscale; higher score = greater severity of symptoms. Negative value = reduction from baseline (b), positive value = increase from b. Change = (HADS score at observation period minus HADS score at b) divided by HADS score b.
Time Frame: Week 21, LOCF
Population: FAS. LOCF = Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 135
scores on scale
  Week 21: Anxiety | -1.4 (3.7)
  LOCF: Anxiety | -1.4 (3.8)
  Week 21: Depression | -0.8 (4.8)
  LOCF: Depression | -0.7 (4.7)
Statistical Analysis 1: Comparison: Pregabalin; Anxiety: Week 21. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Pregabalin; Anxiety: LOCF. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p < .0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Pregabalin; Depression: Week 21. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.0799, t-test, 2 sided
Statistical Analysis 4: Comparison: Pregabalin; Depression: LOCF. Change from baseline evaluated by a one-sample two-sided t-test comparing the difference to zero; Test type: Superiority or Other; p = 0.0846, t-test, 2 sided

ADVERSE EVENTS:
Description: Safety population = all subjects who took at least 1 dose of study medication. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 8/136
Other Adverse Events (participants affected / at risk) | 91/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=136)
Vertigo (Ear and labyrinth disorders) | 2
Drug intolerance (General disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Grand mal convulsion (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Partial seizures with secondary generalization (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=136)
Ear pain (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 7
Conjunctival irritation (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Odynophagia (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Tootheache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Irritability (General disorders) | 1
Pyrexia (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Face injury (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skin injury (Injury, poisoning and procedural complications) | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1
Weight increased (Investigations) | 19
Overweight (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 25
Dysaesthesia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dyslalia (Nervous system disorders) | 1
Head discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 12
Paraesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 59
Tension headache (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agoraphobia (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Spontaneous penile erection (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Scar (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.